CLINICAL TRIAL: NCT03215186
Title: Establishment of the Mathematic Model of Non-genetic Risk Factors of Congenital Cataracts
Brief Title: Non-genetic Risk Factors of Congenital Cataracts
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Home for Cataract Children, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: CCPMOH2017-China-2
Record Dates: First submitted 2017-07-06; First posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Cataract
Keywords: congenital cataract; risk factor; mathematic model
MeSH Terms: conditions — Cataract | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cataract children: All children in this group were diagnosed as congenital cataracts. The four respects of following information of CC patients were collected and confirmed: 1) demography: including age, sex, and laterality; 2) family and pregnancy-labor histories: including family history, mothers' disease and medication histories during pregnancy, premature or term infant, cesarean or eutocia, and history of oxygen inspiration/infant incubator; 3) complicated systemic diseases; 4) living environment: including radiation/pollution exposure, parental smoking, parental education level, and family income.
  Interventions: Other: observational study
- Healthy children: All children in this group were healthy and without cataracts. The four respects of following information of CC patients were collected and confirmed: 1) demography: including age, sex, and laterality; 2) family and pregnancy-labor histories: including family history, mothers' disease and medication histories during pregnancy, premature or term infant, cesarean or eutocia, and history of oxygen inspiration/infant incubator; 3) complicated systemic diseases; 4) living environment: including radiation/pollution exposure, parental smoking, parental education level, and family income.

INTERVENTIONS:
Other: observational study
  Groups: Cataract children

SUMMARY:
Prevention and treatment of the reversible childhood blindness, including congenital cataracts (CC), has been listed as a significant component of the international programme "VISION 2020 - the Right to Sight" launched by WHO in 1999. However, there is still a lot of unsolved problems regarding to CC, especially in developing countries, such as the delayed presentation and treatment to the hospitals, the lack of specialized treatment departments, and the poor treatment prognosis. With the two children policy opened in China in 2016, many CC parents hesitate to have a second child due to the potential high risk of CC. Date on detailed clinical characteristics of the CC children, including the demography, pregnancy-labor history, and living condition, are crucial for developing the national screening strategies of CC in Pregnant women. However, to our knowledge, it still lacks of thus large population-based and comprehensive investigations of the characteristics of CC children in developing countries.

DETAILED DESCRIPTION:
Prevention and treatment of the reversible childhood blindness, including congenital cataracts (CC), has been listed as a significant component of the international programme "VISION 2020 - the Right to Sight" launched by WHO in 1999. However, there is still a lot of unsolved problems regarding to CC, especially in developing countries, such as the delayed presentation and treatment to the hospitals, the lack of specialized treatment departments, and the poor treatment prognosis. With the two children policy opened in China in 2016, many CC parents hesitate to have a second child due to the potential high risk of CC. Date on detailed clinical characteristics of the CC children, including the demography, pregnancy-labor history, and living condition, are crucial for developing the national screening strategies of CC in Pregnant women. However, to our knowledge, it still lacks of thus large population-based and comprehensive investigations of the characteristics of CC children in developing countries. Supporting by the National Ministry of Health and the Zhongshan Ophthalmic Center (ZOC), a specialized eye facility with the largest CC database in China, we therefore comprehensively investigated the demography, pregnancy-labor history, and living condition of CC children with their first visits to the hospital. We also further established a mathematic model of non-genetic risk factors of congenital cataracts. The implications of this study will be of clinical importance to roughly predict the risk of CC in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congenital cataract.
* Less than 18 years old.

Exclusion Criteria:

* The children with definite or suspected ocular trauma (including blunt trauma) history and those with regular ocular or systemic steroid history were excluded from this study.
* The children came from the welfare homes with unclear family heredity and gestation history information were also excluded.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The prospective study included congenital cataract (CC) patients ≤ 18 years old and firstly present to the ZOC in Guangzhou from 2011 to 2017. The included patients registered in the CC database after being diagnosed as CC by at least two experienced pediatric ophthalmologists based on the slit-lamp and Pentacam examinations. The detailed basic information of each CC patient including the demography, family heredity, gestation history, complicated systemic disease, living condition and the family environment were investigated to parents by a structured questionnaire and were recorded in the CC database. The healthy children without CC were set as control. More than 1000 subjects should be included in each group.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-02-01 (Actual); Primary Completion 2018-02-28 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Demography (age, sex, and laterality) | Baseline
  The demography of cataract and healthy children were recorded by using a semi-structured questionnaire.
Family and pregnancy-labor histories (family history, mothers' disease and medication histories during pregnancy, premature or term infant, cesarean or eutocia, and history of oxygen inspiration/infant incubator) | Baseline
  Measured by using a semi-structured questionnaire.
Complicated systemic diseases (congenital heart diseases, brain diseases, favism, etc.) | Baseline
  Measured by using a semi-structured questionnaire.
Living environment (radiation/pollution exposure, parental smoking, parental education) | Baseline
  Measured by using a semi-structured questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D. Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Lin H, Long E, Chen W, Liu Y. Documenting rare disease data in China. Science. 2015 Sep 4;349(6252):1064. doi: 10.1126/science.349.6252.1064-b. No abstract available. PMID 26339020
- See also: Description Description Home page of Zhongshan Ophthalmic Center — http://www.gzzoc.com/